CLINICAL TRIAL: NCT00921349
Title: A Randomized, Controlled Trial of Ligation Plus Nadolol Versus Nadolol Alone in the Prophylaxis of First Variceal Bleeding in Cirrhosis
Brief Title: A Trial of Ligation Plus Nadolol Versus Nadolol Alone in the Prophylaxis of First Variceal Bleeding in Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: National Science Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EVL+Nadolol
Record Dates: First submitted 2009-06-03; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Variceal Bleeding; Cirrhosis
Keywords: Prophylaxis; ligation; beta blockers; First bleeding rate
MeSH Terms: conditions — Fibrosis | interventions — Nadolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ligation+Nadolol (Experimental): Multi-ligators were applied. Patients received regular ligation treatment at an interval of 3-4 weeks until variceal obliteration.
  Intervention; ligation of varices plus beta blockers (Nadolol).
  Interventions: Procedure: Ligation of varices; Drug: Nadolol
- Nadolol only (Active Comparator)
  Interventions: Drug: Nadolol

INTERVENTIONS:
Procedure: Ligation of varices — all varices are ligated until obliteration
  Arms: Ligation+Nadolol
Drug: Nadolol — Nadolol (beta-blocker)

SUMMARY:
The value of banding ligation plus beta blocker in the prophylaxis of first episodes of variceal bleeding has not yet been evaluated. This study was conducted to compare the efficacy and safety of banding ligation plus nadolol versus nadolol in the prophylaxis of first bleeding in cirrhotic patients with high-risk esophageal varices.

DETAILED DESCRIPTION:
Currently, endoscopic variceal ligation (EVL) has replaced EIS as the endoscopic treatment of choice for management of bleeding esophageal varices. The advantages of EVL include requiring fewer treatment sessions to achieve variceal obliteration, lower rebleeding rates and fewer complications (5-9). Controlled studies that compared EVL with beta-blocker in the prevention of first variceal bleeding suggested that EVL was at least equal to beta-blockers in the prophylaxis of first variceal bleeding. However, portal pressure may be elevated after repeated EVL. Hence the combination of nadolol and EVL is a reasonable approach to prevent the first episode of variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. the cause of portal hypertension was cirrhosis
2. the degree of esophageal varices was F2 (moderate varices) or more, associated with any of red color signs (red wale markings, cherry red spots or hematocystic spots)
3. no history of hemorrhage from esophageal varices
4. no current treatment with beta-blockers
5. cirrhosis was based on results of liver biopsy, or clinical and biochemical examinations and image studies

Exclusion Criteria:

1. age greater than 75 years old or younger than 20 years old
2. association with malignancy, uremia or other serious medical illness which may reduce the life expectancy
3. presence of refractory ascites, hepatic encephalopathy or marked jaundice (serum bilirubin > 10 mg/dl)
4. history of shunt operation, transjugular intrahepatic portosystemic stent shunt or endoscopic therapy (EIS or EVL)
5. had contraindications to beta-blockers, such as asthma, heart failure, complete atrioventricular block, hypotension ( systolic blood pressure < 90 mmHg), pulse rate < 60/ min
6. unable to cooperate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary end points of the study were the first episode of variceal bleeding. | 2 years

SECONDARY OUTCOMES:
The secondary end points were adverse events related to treatment and death of any cause. | 2 years